CLINICAL TRIAL: NCT04701905
Title: The Offer of Neurosurgery Care in the Grand Est of France During the Health Crisis Linked to Covid-19
Acronym: NeurochirCOVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7780
Record Dates: First submitted 2021-01-07; First posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: COVID-19 Pandemic
Keywords: COVID-19 Pandemic; Coronavirus; Sars-cov-2
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
During this exceptional health crisis, this study of the current care of a neurosurgical activity, which is essential in a University Hospital Centre, will enable us to better understand how we function, the response given to a population with the means at our disposal, the implementation of new therapeutic strategies and their limits, ethical reflection, and, how to pursue a distributive and quality medicine.

The restriction of conventional medical resources to our care activity (resuscitation, personnel, operating theatre, constraints linked to the risk of contamination...) is leading to a new medical organisation imposing new Covid-19 standards, the description of which seems essential to us.

A knowledge of the strategies to be adopted during a disaster health situation in order to continue providing care to the civilian population. How can we prevent the setting up of health care systems outside the cause of the health crisis? n triage medicine, Avoiding the "burn-out" of doctors struck by the health crisis.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 18;
* Entering the neurosurgery care sector requiring support between 03/16/2020 and 06/15/2020;
* Having not expressed his opposition, after information, to the reuse of his data for the purposes of this research.

Exclusion Criteria:

* Subject having expressed opposition to participating in the study
* Subject under guardianship or guardianship
* Subject under safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient entering the neurosurgery care sector requiring treatment between 03/16/2020 and 06/15/2020
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2020-04-30 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Retrospective analysis of the management of neurosurgical pathologies in a health crisis situation of the Covid-19 pandemic | The files analysed retrospectily from March 16, 2020 to June 15, 2020 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: François PROUST, MD, PhD, Principal Investigator — Department of Neurosurgery - Strasbourg University Hospitals
Locations (1):
- Department of Neurosurgery - Strasbourg University Hospitals, Strasbourg, France